CLINICAL TRIAL: NCT04728971
Title: To Evaluate the Efficacy and Safety of Micafungin in Preventing Invasive Mycosis After Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lin Zhong, Director of Hepatobiliary and Pancreatic Surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHLTQC-4
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Liver Transplantation
Keywords: Micafungin; Invasive Mycosis; Prevention
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Micafungin; Injections; Caspofungin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micafungin Preventing Group (Experimental)
  Interventions: Drug: Micafungin Sodium 50 MG Injection
- Others Preventing Group (Active Comparator)
  Interventions: Drug: Caspofungin Acetate

INTERVENTIONS:
Drug: Micafungin Sodium 50 MG Injection — Give Micafungin 150 mg/d within 24 hours after liver transplantation.
  Arms: Micafungin Preventing Group
Drug: Caspofungin Acetate — Give Caspofungin 35 mg/d lasts 1 week after liver transplantation.
  Arms: Others Preventing Group

SUMMARY:
To evaluate the clinical success rate of micafungin in preventing invasive mycosis after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily;
2. Liver transplant patients with 1 high-risk factor; A. Transplant again; B. Fulminant liver failure; C. Renal failure requires alternative treatment (defined as creatinine clearance ≤40 ml/min); D. ICU duration before liver transplantation≥48h; E. Have received abdominal surgery within one month before liver transplantation or; F. Common bile duct jejunostomy (except for children); G. Excessive blood transfusion (blood transfusion exceeds 2000mL); H. The donor's ICU hospital stay exceeds 5 days; I. Positive sputum and blood culture of the donor J. The donor has evidence of lung or bloodstream infection (pulmonary infection is evaluated according to the diagnostic criteria and treatment principles (draft) of invasive lung fungal infection, and bloodstream infection is evaluated according to invasive fungal disease of patients with hematopathy/malignant tumor Diagnostic criteria and treatment principles (fifth revised edition) for evaluation) K. 60 years old ≤ age ≤ 65 years old

Exclusion Criteria:

1. Have used other investigational drugs or are participating in other clinical trials within 4 weeks before enrollment;
2. Currently combined with any kind of fungal infection;
3. Allergic to study drugs;
4. Joint transplantation;
5. Women who are pregnant, preparing to become pregnant or breast-feeding;
6. The investigator thinks that it is not suitable to use the test drug.

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Post-transplant infections | 90 days
  Frequency of clinically or microbiologically documented infection after transplantation.